CLINICAL TRIAL: NCT06889103
Title: Psychometric Properties of the Turkish Version of the Edinburgh Feeding Evaluation in Dementia (EdFed) Scale
Brief Title: Turkish Edinburgh Feeding Evaluation in Dementia (EdFed) Scale
Acronym: EdFed
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Busra Kul, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: Edfed scale
Record Dates: First submitted 2025-01-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Feeding Difficulties; Reliability and Validity
Keywords: dementia; EdFed; interobserver agreement
MeSH Terms: conditions — Dementia | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observed: observation during eating
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — observation during eating

SUMMARY:
This study was conducted to evaluate the psychometric properties, including interobserver agreement, of the Turkish version of the Edinburgh Feeding Evaluation in Dementia (EdFed) scale, which was developed to assess eating difficulties in patients with dementia.

DETAILED DESCRIPTION:
Eating difficulties are common in dementia patients and can lead to malnutrition. Early detection and intervention of these difficulties is of great importance to minimise the negative effects. Therefore, a reliable and valid tool for assessing nutritional difficulties in dementia patients is needed.

ELIGIBILITY:
Inclusion Criteria:

* Those over the age of 65,
* Those diagnosed with dementia,
* Patients who are able to weigh themselves (no lower extremity loss)

Exclusion Criteria:

• (CDR<2)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Nursing home
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Edfed score | 1 year
  Psychometric properties of the Turkish version of the Edinburgh Feeding Evaluation in Dementia (EdFed) scale

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Kul, MsC, Principal Investigator — ÜSKÜDAR ÜNİVERSİTESİ; Zelıha Tulek, Proffessor, Study Director — İstanbul University-Cerrahpaşa
Locations (1):
- Darülaceze, Istanbul, Sıslı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It can be shared after publication.

REFERENCES:
- [Background] Bagnasco A, Watson R, Zanini M, Rosa F, Rocco G, Sasso L. Preliminary testing using Mokken scaling of an Italian translation of the Edinburgh Feeding Evaluation in Dementia (EdFED-I) scale. Appl Nurs Res. 2015 Nov;28(4):391-6. doi: 10.1016/j.apnr.2015.02.003. Epub 2015 Feb 26. PMID 26608444